CLINICAL TRIAL: NCT00532896
Title: Impact of Weight Loss Following Bariatric Surgery on Pulmonary Function in Patients With Morbid Obesity
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Louis-Philippe Boulet, MD, FRCPC, FCCP, Laval University
Other Study IDs: HL-Ch-BAR-Pneu-20086
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Bariatric Surgery; Obesity; Respiratory Diseases
MeSH Terms: conditions — Obesity; Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- bariatric surgery: patients with morbid obesity undergoing a bariatric surgery
- No bariatric surgery: patients with morbid obesity on a waiting list for a bariatric surgery but who will have their surgery in more than one year.

SUMMARY:
Increase in body mass index (BMI)is associated with a decrease in expiratory flows.Obesity is also associated with an increased prevalence of asthma.Consequences of obesity on respiratory function and on bronchial responsiveness are still to be documented.

This study aims to evaluate, before and after surgery, the impact of a bariatric surgery (biliopancreatic diversion with duodenal switch)on respiratory function in patients with morbid obesity .

Our hypothesis is that weight loss following bariatric surgery will induce significant improvements in pulmonary function and airway responsiveness, and, as a consequence, a reduction in respiratory symptoms,these changes being correlated with a reduction in systemic markers of inflammation. Maintenance of weight loss after one year will permit the persistence of these improvements

DETAILED DESCRIPTION:
Patients will be evaluated before the surgery (time zero), 6 months and one year after their surgery. A control group of patients on a waiting list for bariatric surgery will be evaluated at time zero and after 6 months and one year.

At each visit,patients will:

* fill a standardized respiratory questionnaire and a questionnaire on sleep apnea; questionnaires on asthma control will be completed by patients with asthma.
* have a spirometry, pulmonary volumes measures by body plethysmography and methacholine inhalation test with evaluation of symptoms perception.
* an induced sputum will be performed.
* A blood sample will be drawn to evaluate inflammation and measure C-reactive protein concentration in plasma.
* An allergy skin prick test will be done at time zero.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index >or= 35 kg/m2
* Non-smokers or ex-smokers (<10 packs-year)

Exclusion Criteria:

* Previous bariatric surgery
* previous vagotomy
* no compliance to visits
* subjects unable to provide an informed consent or to understand the questions included in questionnaires
* Patients with cardiac pacemaker
* hemodynamically significant valvulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects on the waiting list for bariatric surgery at Laval Hospital will be offered to participate to the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2006-04; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, Principal Investigator — Hôpital Laval
Locations (1):
- Centre de Recherche, Hôpital Laval, Québec, Quebec, Canada

REFERENCES:
- [Derived] Boulet LP, Turcotte H, Martin J, Poirier P. Effect of bariatric surgery on airway response and lung function in obese subjects with asthma. Respir Med. 2012 May;106(5):651-60. doi: 10.1016/j.rmed.2011.12.012. Epub 2012 Feb 10. PMID 22326605